CLINICAL TRIAL: NCT00968812
Title: A Randomized, Double-Blind, 3-Arm Parallel-Group, 2-Year (104-Week), Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-28431754 Compared With Glimepiride in the Treatment of Subjects With Type 2 Diabetes Mellitus Not Optimally Controlled on Metformin Monotherapy
Brief Title: CANagliflozin Treatment And Trial Analysis-Sulfonylurea (CANTATA-SU) SGLT2 Add-on to Metformin Versus Glimepiride
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016480; 28431754DIA3009 (Other: Janssen Research & Development, LLC); 2009-009320-36 (EudraCT Number)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Metformin; Glimepiride; Hemoglobin A1c; Type 2 diabetes mellitus; Canagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — glimepiride; Sulfonylurea Compounds; Canagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glimepiride (Active Comparator): Each patient will receive glimepiride, at protocol-specified doses, once daily in combination with protocol-specified doses of metformin for 104 weeks.
  Interventions: Drug: Glimepiride; Drug: Metformin
- Canagliflozin 100 mg (Experimental): Each patient will receive 100 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Metformin
- Canagliflozin 300 mg (Experimental): Each volunteer will receive 300 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Metformin

INTERVENTIONS:
Drug: Glimepiride — Glimepiride will be given orally (by mouth), as over-encapsulated tablets, starting at a dose of 1mg once daily and increasing to a maximum of 6 mg or 8 mg once daily for 104 weeks.
  Other Names: sulfonylurea
  Arms: Glimepiride
Drug: Canagliflozin (JNJ-28431754) — Canagliflozin (JNJ-28431754) will be given orally as over-encapsulated tablets, at a dose of 100 mg or 300 mg once daily for 104 weeks.
  Arms: Canagliflozin 100 mg; Canagliflozin 300 mg
Drug: Metformin — Metformin will be given orally at the protocol-specified dose for 104 weeks.

SUMMARY:
The purpose of this study is to demonstrate the efficacy, safety, and tolerability of canagliflozin (JNJ-28431754) compared with glimepiride in patients with type 2 diabetes mellitus with inadequate control despite treatment with metformin.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is well recognized as a major public health problem that presents patients with a significant risk of complications including heart disease, retinopathy, nephropathy, and neuropathy. Various classes of orally administered antihyperglycemic agents have been developed for the treatment of diabetes and although individual agents may be highly effective for some patients, it is still difficult to maintain optimal glycemic control in most patients, thereby resulting in high rates of morbidity and mortality in the diabetic population. This is a randomized, double-blind, active comparator-controlled, 3-arm, parallel-group, multicenter study to demonstrate the efficacy, safety, and tolerability of canagliflozin compared with a sulfonylurea (glimepiride) in patients with T2DM, 18 to 80 years of age, inclusive, who are not optimally controlled on metformin monotherapy. The primary study hypothesis is that the study drug will be non-inferior to glimepiride as assessed by the change in hemoglobin A1c (HbA1c) from baseline. The patients will receive capsules taken by mouth of canagliflozin (either 100 or 300 mg), or glimepiride with a starting dosage of 1 mg, which will be increased to a maximum dose of 6 or 8 mg once daily for a total duration of 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of type 2 diabetes
* Body mass index (BMI) >=22 to <=45 kg/m2, at screening
* Patients must be taking a stable dosage of metformin as monotherapy at screening
* Patients must have a HbA1c between >=7% and <=9.5% at Week 2
* Patients must have a fasting plasma glucose (FPG) <=270 mg/dL (15 mmol/L) at Week -2

Exclusion Criteria:

* Patients having prior exposure or known contraindication or suspected hypersensitivity to JNJ-28431754, glimepiride, or metformin
* History of diabetic ketoacidosis or type 1 diabetes mellitus
* History of pancreas or beta-cell transplantation
* History of active proliferative diabetic retinopathy
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria
* Renal disease requiring treatment with immunosuppressive therapy within the past 12 months before screening or a history of dialysis or renal transplant
* Taken thiazolidinedione therapy in the past 16 weeks before screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1452 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (138):
- United States (43):
  - Calera, Alabama
  - Gilbert, Arizona
  - Mesa, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Buena Park, California
  - Encinitas, California
  - Fresno, California
  - Lincoln, California
  - Roseville, California
  - San Diego, California
  - Westlake Village, California
  - Chipley, Florida
  - Marianna, Florida
  - Oldsmar, Florida
  - Orlando, Florida
  - Augusta, Georgia
  - Perry, Georgia
  - Nampa, Idaho
  - Chicago, Illinois
  - Vernon Hills, Illinois
  - Valparaiso, Indiana
  - New Orleans, Louisiana
  - Elkridge, Maryland
  - Bloomfield Hills, Michigan
  - Las Vegas, Nevada
  - Canal Fulton, Ohio
  - Gallipolis, Ohio
  - Mason, Ohio
  - Perrysburg, Ohio
  - Tulsa, Oklahoma
  - Yukon, Oklahoma
  - Fleetwood, Pennsylvania
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Odessa, Texas
  - Pearland, Texas
  - San Antonio, Texas
  - Danville, Virginia
  - Olympia, Washington
  - Milwaukee, Wisconsin
  - Wauwatosa, Wisconsin
- Argentina (3):
  - Buenos Aires
  - Mar del Plata
  - Rosario
- Bulgaria (4):
  - Dimitrovgrad
  - Kazanlak
  - Rousse
  - Sofia
- Canada (8):
  - Chilliwack, British Columbia
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Mississauga, Ontario
  - Toronto, Ontario
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- Costa Rica (2):
  - San José
  - San Pedro
- Denmark (4):
  - Aalborg
  - Ballerup Municipality
  - Vejle
  - Vipperoed
- Finland (5):
  - Helsinki
  - Kokkola
  - Kuopio
  - Oulu
  - Turku
- Germany (6):
  - Berlin
  - Dresden
  - Düsseldorf
  - Hamburg
  - Mainz
  - Villingen-Schwenningen
- India (7):
  - Bangalore
  - Chennai
  - Coimbatore
  - Hyderabad
  - Nagpur
  - Pune
  - Wardha
- Israel (8):
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Ramat Gan
  - Rehovot
  - Safed
  - Tel Aviv
- Mexico (3):
  - Mexico City
  - México
  - Monterrey
- Norway (2):
  - Ålesund
  - Oslo
- Philippines (4):
  - Cebu
  - Marikina City
  - Pasay
  - Quezon City
- Poland (9):
  - Bydgoszcz
  - Krakow
  - Kutno
  - Lodz
  - Lublin
  - Torun
  - Warsaw
  - Wroclaw
  - Zielona Góra
- Ponce, Puerto Rico
- Romania (7):
  - Baia Mare
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Galati
  - Ploieşti
  - Târgu Mureş
- Russia (5):
  - Arkhangelsk
  - Moscow
  - Saint Petersburg
  - Samara
  - Saratov
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Ľubochňa
  - Prešov
- South Korea (7):
  - Daegu
  - Goyang-si
  - Gyeonggi-do
  - Incheon
  - Seoul
  - Suwon
  - Wŏnju
- Ukraine (6):
  - Dnipro
  - Kharkiv
  - Kiev
  - Poltava
  - Ternopil
  - Vinnitsa

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Heerspink HJL, Perco P, Mulder S, Leierer J, Hansen MK, Heinzel A, Mayer G. Canagliflozin reduces inflammation and fibrosis biomarkers: a potential mechanism of action for beneficial effects of SGLT2 inhibitors in diabetic kidney disease. Diabetologia. 2019 Jul;62(7):1154-1166. doi: 10.1007/s00125-019-4859-4. Epub 2019 Apr 17. PMID 31001673
- [Derived] Garvey WT, Van Gaal L, Leiter LA, Vijapurkar U, List J, Cuddihy R, Ren J, Davies MJ. Effects of canagliflozin versus glimepiride on adipokines and inflammatory biomarkers in type 2 diabetes. Metabolism. 2018 Aug;85:32-37. doi: 10.1016/j.metabol.2018.02.002. Epub 2018 Feb 13. PMID 29452178
- [Derived] Qiu R, Balis D, Xie J, Davies MJ, Desai M, Meininger G. Longer-term safety and tolerability of canagliflozin in patients with type 2 diabetes: a pooled analysis. Curr Med Res Opin. 2017 Mar;33(3):553-562. doi: 10.1080/03007995.2016.1271780. Epub 2017 Jan 4. PMID 27977934
- [Derived] John M, Cerdas S, Violante R, Deerochanawong C, Hassanein M, Slee A, Canovatchel W, Hamilton G. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus living in hot climates. Int J Clin Pract. 2016 Sep;70(9):775-85. doi: 10.1111/ijcp.12868. PMID 27600862
- [Derived] Patel CA, Bailey RA, Vijapurkar U, Meininger G, Blonde L. A post-hoc analysis of the comparative efficacy of canagliflozin and glimepiride in the attainment of type 2 diabetes-related quality measures. BMC Health Serv Res. 2016 Aug 5;16(a):356. doi: 10.1186/s12913-016-1607-z. PMID 27495291
- [Derived] Blonde L, Stenlof K, Fung A, Xie J, Canovatchel W, Meininger G. Effects of canagliflozin on body weight and body composition in patients with type 2 diabetes over 104 weeks. Postgrad Med. 2016 May;128(4):371-80. doi: 10.1080/00325481.2016.1169894. Epub 2016 Apr 7. PMID 27002421
- [Derived] Leiter LA, Langslet G, Vijapurkar U, Davies MJ, Canovatchel W. Simultaneous Reduction in Both HbA1c and Body Weight with Canagliflozin Versus Glimepiride in Patients with Type 2 Diabetes on Metformin. Diabetes Ther. 2016 Jun;7(2):269-78. doi: 10.1007/s13300-016-0163-1. Epub 2016 Mar 16. PMID 26984361
- [Derived] Watts NB, Bilezikian JP, Usiskin K, Edwards R, Desai M, Law G, Meininger G. Effects of Canagliflozin on Fracture Risk in Patients With Type 2 Diabetes Mellitus. J Clin Endocrinol Metab. 2016 Jan;101(1):157-66. doi: 10.1210/jc.2015-3167. Epub 2015 Nov 18. PMID 26580237
- [Derived] Lavalle-Gonzalez FJ, Eliaschewitz FG, Cerdas S, Chacon Mdel P, Tong C, Alba M. Efficacy and safety of canagliflozin in patients with type 2 diabetes mellitus from Latin America. Curr Med Res Opin. 2016;32(3):427-39. doi: 10.1185/03007995.2015.1121865. Epub 2016 Jan 14. PMID 26579834
- [Derived] Leiter LA, Yoon KH, Arias P, Langslet G, Xie J, Balis DA, Millington D, Vercruysse F, Canovatchel W, Meininger G. Canagliflozin provides durable glycemic improvements and body weight reduction over 104 weeks versus glimepiride in patients with type 2 diabetes on metformin: a randomized, double-blind, phase 3 study. Diabetes Care. 2015 Mar;38(3):355-64. doi: 10.2337/dc13-2762. Epub 2014 Sep 9. PMID 25205142
- [Derived] Nyirjesy P, Sobel JD, Fung A, Mayer C, Capuano G, Ways K, Usiskin K. Genital mycotic infections with canagliflozin, a sodium glucose co-transporter 2 inhibitor, in patients with type 2 diabetes mellitus: a pooled analysis of clinical studies. Curr Med Res Opin. 2014 Jun;30(6):1109-19. doi: 10.1185/03007995.2014.890925. Epub 2014 Feb 21. PMID 24517339
- [Derived] Cefalu WT, Leiter LA, Yoon KH, Arias P, Niskanen L, Xie J, Balis DA, Canovatchel W, Meininger G. Efficacy and safety of canagliflozin versus glimepiride in patients with type 2 diabetes inadequately controlled with metformin (CANTATA-SU): 52 week results from a randomised, double-blind, phase 3 non-inferiority trial. Lancet. 2013 Sep 14;382(9896):941-50. doi: 10.1016/S0140-6736(13)60683-2. Epub 2013 Jul 12. PMID 23850055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin (JNJ-28431754) compared with glimepiride in participants with type 2 diabetes mellitus with inadequate glycemic control despite metformin treatment. The study was conducted between 28 August 2009 and 25 January 2013 and included 157 study centers in 19 countries worldwide.
Pre-assignment Details: 1,452 participants were randomly allocated to the 3 treatment arms. 1450 participants received at least 1 dose of study drug and were included in the modified intent-to-treat (mITT) analysis set and safety analysis set. Participant flow is presented for Baseline to Week 104.
Groups:
- Canagliflozin 100 mg: Baseline to Week 104: Each patient received 100 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks.
- Canagliflozin 300 mg: Baseline to Week 104: Each patient received 300 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks.
- Glimepiride: Baseline to Week 104: Each patient received glimepiride, at protocol-specified doses, once daily in combination with protocol-specified doses of metformin for 104 weeks.
Period: Overall Study
Arm/Group | Canagliflozin 100 mg: Baseline to Week 104 | Canagliflozin 300 mg: Baseline to Week 104 | Glimepiride: Baseline to Week 104
Started | 483 | 485 | 482
Completed | 343 | 323 | 314
Not Completed | 140 | 162 | 168
Not completed — Adverse Event | 30 | 46 | 33
Not completed — Death | 2 | 2 | 1
Not completed — Lack of Efficacy | 9 | 7 | 16
Not completed — Lost to Follow-up | 17 | 12 | 11
Not completed — Physician Decision | 8 | 5 | 9
Not completed — Protocol Violation | 7 | 4 | 3
Not completed — Withdrawal by Subject | 17 | 23 | 25
Not completed — Creatinine or eGFR withdrawal criteria | 9 | 13 | 7
Not completed — Noncompliance with study drug | 4 | 1 | 6
Not completed — Unable to take rescue therapy | 12 | 12 | 17
Not completed — Other | 25 | 37 | 40

BASELINE CHARACTERISTICS:
Groups:
- Canagliflozin 100 mg: Each patient received 100 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks.
- Canagliflozin 300 mg: Each patient received 300 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks.
- Glimepiride: Each patient received glimepiride, at protocol-specified doses, once daily in combination with protocol-specified doses of metformin for 104 weeks.
- Total: Total of all reporting groups
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Glimepiride | Total
Number analyzed (Participants) | 483 | 485 | 482 | 1450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 397 | 411 | 399 | 1207
  >=65 years | 86 | 74 | 83 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.49) | 55.8 (9.17) | 56.3 (9.01) | 56.2 (9.22)
Gender [Count of Participants; unit: Participants]
  Female | 231 | 244 | 219 | 694
  Male | 252 | 241 | 263 | 756
Region Enroll [Number; unit: participants]
  ARGENTINA | 18 | 18 | 18 | 54
  BULGARIA | 7 | 7 | 7 | 21
  CANADA | 19 | 20 | 19 | 58
  COSTA RICA | 10 | 9 | 9 | 28
  DENMARK | 24 | 25 | 25 | 74
  FINLAND | 18 | 17 | 19 | 54
  GERMANY | 6 | 7 | 6 | 19
  INDIA | 55 | 55 | 56 | 166
  ISRAEL | 14 | 15 | 14 | 43
  MEXICO | 24 | 25 | 24 | 73
  NORWAY | 9 | 9 | 9 | 27
  PHILIPPINES | 14 | 13 | 13 | 40
  POLAND | 14 | 15 | 15 | 44
  ROMANIA | 43 | 43 | 44 | 130
  RUSSIAN FEDERATION | 23 | 22 | 22 | 67
  SLOVAKIA | 15 | 14 | 13 | 42
  SOUTH KOREA | 31 | 32 | 31 | 94
  UKRAINE | 22 | 22 | 22 | 66
  UNITED STATES | 117 | 117 | 116 | 350

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 52 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus glimepiride) in the LS mean change.
Time Frame: Day 1 (Baseline) and Week 52
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug). Last-observation-carried-forward method used for missing Week 52 values. Measurements taken pre-rescue used as last observation in patients receiving glycemic rescue therapy. Table includes only patients with both baseline and post baseline values.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Glimepiride
Number analyzed (Participants) | 478 | 474 | 473
Percent | -0.82 (0.039) | -0.93 (0.039) | -0.81 (0.039)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Glimepiride; If the hypothesis of non-inferiority of canagliflozin to glimepiride at Week 52 was demonstrated (ie, upper bound of the 95% Confidence Interval of the treatment difference [canagliflozin minus glimepiride] was less than 0.3) and the upper bound was less than 0.0, the superiority of the canagliflozin dose relative to glimepiride would be concluded; Test type: Non-Inferiority or Equivalence — Power calculation: assuming a difference between canagliflozin and glimepiride of 0.0% and a common standard deviation of 1.0%, and using a 2-sample, 1-sided t-test with a Type I error rate of 0.0125, and assuming a drop-out rate of 35% in 52 weeks, it was estimated that approximately 427 patients per group would provide 90% power to demonstrate non-inferiority with the non-inferiority margin of 0.3, comparing canagliflozin with glimepiride; ANCOVA; Least-Squares Mean Difference = -0.01, 95% CI 2-sided [-0.109 to 0.085], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Least-Squares Mean Difference = -0.12, 95% CI 2-sided [-0.217 to -0.023], Standard Error of Mean 0.050

2. Secondary Outcome: Percentage of Patients Experiencing at Least 1 Hypoglycemic Event From Baseline to Week 52
Description: The table below shows the percentage of patients who experienced at least 1 documented hypoglycemic event from Baseline to Week 52 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus glimepiride) in percentages.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Glimepiride
Number analyzed (Participants) | 483 | 485 | 482
Percentage of patients | 5.6 | 4.9 | 34.2
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Glimepiride; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.06 to 0.16]
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Glimepiride; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.09, 95% CI 2-sided [0.05 to 0.14]

3. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 52
Description: The table below shows the least-squares (LS) mean percent change in body weight from Baseline to Week 52 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus glimepiride) in the LS mean percent change.
Time Frame: Day 1 (Baseline) and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Glimepiride
Number analyzed (Participants) | 479 | 480 | 478
Percent change | -4.2 (0.2) | -4.7 (0.2) | 1.0 (0.2)
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -5.2, 95% CI 2-sided [-5.7 to -4.7], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Least-Squares Mean Difference = -5.7, 95% CI 2-sided [-6.2 to -5.1], Standard Error of Mean 0.3

4. Secondary Outcome: Change in HbA1c From Baseline to Week 104
Description: The table below shows the least-squares (LS) mean change in HbA1c from Baseline to Week 104 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin group minus glimepiride) in the LS mean change.
Time Frame: Baseline, Week 104
Population: Analysis used mITT analysis set (all randomized patients who received at least 1 dose of study drug).
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Canagliflozin 100 mg | Canagliflozin 300 mg | Glimepiride
Number analyzed (Participants) | 478 | 474 | 474
Percent | -0.65 (0.042) [0.10 to 0.22] | -0.74 (0.042) [0.10 to 0.21] | -0.55 (0.043) [0.31 to 0.43]
Statistical Analysis 1: Comparison: Canagliflozin 100 mg vs Glimepiride; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = -0.09, 95% CI 2-sided [-0.200 to 0.010], Standard Error of Mean 0.054
Statistical Analysis 2: Comparison: Canagliflozin 300 mg vs Glimepiride; Test type: Superiority or Other; ANCOVA; Least-Squares Mean Difference = -0.18, 95% CI 2-sided [-0.289 to -0.078], Standard Error of Mean 0.054

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study (104 weeks).
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
  MEDDRA 14.1 used for Week 52 / MEDDRA 15.0 for Week 104 results.
Groups:
- Canagliflozin 100 mg: Baseline to Week 52: Each patient received 100 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks. Data are presented for Baseline to Week 52.
- Canagliflozin 300 mg: Baseline to Week 52: Each patient received 300 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks. Data are presented for Baseline to Week 52.
- Glimepiride: Baseline to Week 52: Each patient received glimepiride, at protocol-specified doses, once daily in combination with protocol-specified doses of metformin for 104 weeks. Data are presented for Baseline to Week 52.
- Canagliflozin 100 mg: Baseline to Week 104: Each patient received 100 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks. Data are presented for Baseline to Week 104.
- Canagliflozin 300 mg: Baseline to Week 104: Each patient received 300 mg of canagliflozin (JNJ-28431754) once daily with protocol-specified doses of metformin for 104 weeks. Data are presented for Baseline to Week 104.
- Glimepiride: Baseline to Week 104: Each patient received glimepiride, at protocol-specified doses, once daily in combination with protocol-specified doses of metformin for 104 weeks. Data are presented for Baseline to Week 104.
Arm/Group | Canagliflozin 100 mg: Baseline to Week 52 | Canagliflozin 300 mg: Baseline to Week 52 | Glimepiride: Baseline to Week 52 | Canagliflozin 100 mg: Baseline to Week 104 | Canagliflozin 300 mg: Baseline to Week 104 | Glimepiride: Baseline to Week 104
Serious Adverse Events (participants affected / at risk) | 24/483 | 26/485 | 39/482 | 47/483 | 47/485 | 69/482
Other Adverse Events (participants affected / at risk) | 138/483 | 150/485 | 175/482 | 198/483 | 204/485 | 242/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Canagliflozin 100 mg: Baseline to Week 52 (N=483) | Canagliflozin 300 mg: Baseline to Week 52 (N=485) | Glimepiride: Baseline to Week 52 (N=482) | Canagliflozin 100 mg: Baseline to Week 104 (N=483) | Canagliflozin 300 mg: Baseline to Week 104 (N=485) | Glimepiride: Baseline to Week 104 (N=482)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 2 | 3 | 2 | 3
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 2
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 2
Diabetic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 2 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — This event was re-coded as "Small bowel perforation"; it was subsequently re-mapped to the "Surgical and medical procedures".
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 2 | 0 | 2 | 3
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 0 | 4
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2
Endometritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 — In the Week 52 study report, this event was coded as "infection"; it was subsequently re-coded in the Week 104 study report as "localised infection".
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 1 | 2 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 3 | 0
Carotid arterial embolus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0 | 2 | 1 | 2
Hemiplegic migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — In the Week 52 study report, this event was coded as "Hemiplegic migraine"; it was subsequently re-coded in the Week 104 study report as "Hemiparesis".
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 — In the Week 52 study report, this event was coded as "stress"; it was subsequently re-coded in the Week 104 study report as "anxiety".
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 1 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Philmosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal strangulated herina (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram T wave biphasic (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Complex regional pain syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 — In the Week 52 study report, this event was coded as "Hemiplegic migraine"; it was subsequently re-coded in the Week 104 study report as "Hemiparesis".
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 — In the Week 52 study report, this event was coded as "stress"; it was subsequently re-coded in the Week 104 study report as "anxiety".
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Familial risk factor (Social circumstances) | 0 | 0 | 0 | 0/482 | 1/483 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — In the Week 52 study report, this event was coded as "infection"; it was subsequently re-coded in the Week 104 study report as "localised infection".
Small bowel perforation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 — In Week 52 study report this event was coded as "small intestinal perforation" and was mapped under "Gastrointestinal disorders ".
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Canagliflozin 100 mg: Baseline to Week 52 (N=483) | Canagliflozin 300 mg: Baseline to Week 52 (N=485) | Glimepiride: Baseline to Week 52 (N=482) | Canagliflozin 100 mg: Baseline to Week 104 (N=483) | Canagliflozin 300 mg: Baseline to Week 104 (N=485) | Glimepiride: Baseline to Week 104 (N=482)
Diarrhoea (Gastrointestinal disorders) | 24 | 33 | 29 | 25/482 | 39 | 34
Nausea (Gastrointestinal disorders) | 16 | 25 | 13 | 20 | 27 | 19
Nasopharyngitis (Infections and infestations) | 33 | 37 | 37 | 47 | 55 | 51
Upper respiratory tract infection (Infections and infestations) | 17 | 27 | 41 | 36 | 38 | 56
Urinary tract infection (Infections and infestations) | 26 | 23 | 18 | 44 | 33 | 27
Hypoglycaemia (Metabolism and nutrition disorders) | 15 | 9 | 61 | 17 | 16 | 86
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 18 | 20 | 34 | 28 | 26
Headache (Nervous system disorders) | 14 | 25 | 24 | 21 | 29 | 33
Hypertension (Vascular disorders) | 8 | 10 | 13 | 15 | 11 | 30
Influenza (Infections and infestations) | 14 | 17 | 7 | 25 | 23 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 13 | 18 | 26 | 16 | 24

LIMITATIONS AND CAVEATS:
No notable study limitations were identified by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.